CLINICAL TRIAL: NCT02505256
Title: Study Into Treatment of Hyperplasia of Mammary Glands
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yu-Zhi Gang, Chief of Department of Breast Surgery, Shandong University
Other Study IDs: BEST P-01
Record Dates: First submitted 2015-07-18; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Hyperplasia
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — breast tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- case group: cases who presented as breast pain or breast lumps, and no intervention will be administered.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Hyperplasia of Mammary Glands is a complex disease, and there is no consensus or guideline for the treatment of this disease. This study was launched to investigate into the problem that which patients should be diagnosed as hyperplasia of mammary glands and which patients should be treated.

DETAILED DESCRIPTION:
Females who meet the inclusion criteria will receive breast ultrasonography, mammography and pathological examinations by core needle biopsy. All participants will receive a follow-up at an 6-month interval for 2 years. During the follow-up period, whether the symptoms relieve will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Reported breast pain or breast lumps.
* Willing to be kept follow-up.
* Functions below are maintained in major organs: liver, renal and heart.
* Written informed consent will be obtained for patients for entering this study.

Exclusion Criteria:

* Typical breast cancer or fibroadenoma.
* Classification by breast ultrasonography of mammography is beyond Breast Imaging - Reporting And Data System (BI-RADS) 4.
* Oral contraceptive or hormone replacement therapy.
* History of breast cancer or other malignancies.
* History of pituitary gland disease.
* Potentially pregnant, pregnant, or breast-feeding.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females who reported breast pain of breast lumps.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical manifestations as an substitutive indicator for pathological diagnosis of hyperplasia of mammary glands | 8 months

SECONDARY OUTCOMES:
Clinical manifestations as an surgical indications for hyperplasia of mammary glands | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Gang Z Yu, PhD，MD, Principal Investigator — The Second Hospital of Shandong University
Locations (1):
- the Second Hospital of Shandong Universtity, Jinan, Shandong, China